CLINICAL TRIAL: NCT02199132
Title: Retrospective Study About Nasopharyngeal Carcinoma at C. S. Parc Tauli
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Yolanda Escamilla-Carpintero, MD Phd, Corporacion Parc Tauli
Other Study IDs: CPT_ORL14_YE1
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nasopharyngeal Carcinoma

SUMMARY:
Retrospective study of patients diagnosed with a nasopharyngeal carcinoma included in our data base care between June 1990 and September 2013.

Our hypothesis is:

Our series of patients with a history of nasopharyngeal carcinoma presents epidemiological, response rates to the different treatments and survival similar to those described in the literature

DETAILED DESCRIPTION:
Retrospective study of 50 patients diagnosed with nasopharyngeal carcinoma. The following variables will be studied: age, sex, toxic habits , associated pathology, patient origin , first symptom , duration , histology, stage , second malignancies , recurrences , metastases , treatments performed , the response thereto and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of Nasopharyngeal Carcinoma at Ear-Nose-Throat Department at Corporació Sanitària Parc Taulí from 1993 to 2013

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed of Nasopharyngeal Carcinoma at Ear-Nose-Throught Department at Corporació Sanitària Parc Taulí from 1993 to 2013
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Description of Nasopharyngeal Carcinoma Patients | 1 year after diagnostic
  Describe our population diagnosed nasopharyngeal carcinoma and compared in epidemiology and therapeutic results with those in the literature

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain